CLINICAL TRIAL: NCT00554450
Title: The Pharmacodynamics, Pharmacokinetics, and Safety of Dapagliflozin in Type 2 Diabetic Subjects With Mild, Moderate, and Severe Renal Impairment
Brief Title: Renal Impairment in Type 2 Diabetic Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB102-007
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): 50 mg single dose
  Interventions: Drug: Dapagliflozin
- Arm 2 (Experimental): 20 mg up to 7 days
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, once daily

SUMMARY:
The purpose of the study is to assess the effect of dapagliflozin on renal glucose clearance in type 2 diabetic subjects with mild, moderate, and severe renal impairment compared to type 2 diabetic and healthy subjects with normal renal function

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects in the following groups:

Group A: Healthy Subjects with Normal Renal Function (CLcr > 80 mL/min) Group B: Diabetic Subjects with Normal Renal Function (CLcr > 80 mL/min) Group C: Diabetic Subjects with Mild Renal Impairment (CLcr > 50 - ≤80 mL/min) Group D: Diabetic Subjects with Moderate Renal Impairment (CLcr ≥ 30 - ≤50 mL/min) Group E: Diabetic Subjects with Severe Renal Impairment (CLcr < 30 mL/min) (and not receiving dialysis)

* Men and WOCBP, ages 18 to 79 years old

Standard Exclusion Criteria, plus:

* History of diabetic ketoacidosis
* HbA*1c > 10%
* Serum albumin < 2.0 gm/dL
* Potassium < 3.0 or > 6.0 mEq/L

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Urine will be collected over a 24 h period for determination of renal glucose clearance, total protein, and measurement of total glucose excreted in urine | on Days -1, 1, 4 and 10
Blood samples for serum glucose and creatinine will be collected | on Days -1, 1, 4 and 10 at selected timepoints
Blood and urine PK samples | on Days 1, 4, 10
Iohexol PK blood & urine samples for GFR assessment | on Day -12 to -5

SECONDARY OUTCOMES:
AEs, vital signs | scr, Days -1, 1, 4-11, discharge
physical exams | scr, Days -12 to -5, -1, discharge
ECGs | scr, Days,-1, 4, 7, discharge
clinical labs | scr, Day -1, 1, 4, 6, 8, 10, discharge
The following urine/serum safety parameters will be assessed: sodium, potassium, magnesium, phosphorus, calcium, and total protein (urine only) | on Days -1, 1, 4 and 10

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - Advanced Clinical Research Institute, Anaheim, California
  - Elite Research Institute, Miami, Florida
  - Prism Research, Saint Paul, Minnesota
  - Dgd Research, Inc., San Antonio, Texas

REFERENCES:
- [Result] Kasichayanula S, Liu X, Pe Benito M, Yao M, Pfister M, LaCreta FP, Humphreys WG, Boulton DW. The influence of kidney function on dapagliflozin exposure, metabolism and pharmacodynamics in healthy subjects and in patients with type 2 diabetes mellitus. Br J Clin Pharmacol. 2013 Sep;76(3):432-44. doi: 10.1111/bcp.12056. PMID 23210765
- See also: MB102007 _Redacted _CSR _synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3631&filename=MB102007%20_Redacted%20_CSR%20_synopsis.pdf